CLINICAL TRIAL: NCT00660842
Title: Weekly Versus Every 3 Week Carboplatin and Paclitaxel in Patients With Ovarian Cancer: a Phase III Randomized Multicenter Study
Brief Title: Study Comparing Weekly Versus Every 3 Week Chemotherapy in Patients With Ovarian Cancer
Acronym: MITO-7
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MITO-7; 2008-001754-40 (EudraCT Number)
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cancer
Keywords: quality of life; weekly therapy; neurotoxicity
MeSH Terms: conditions — Ovarian Neoplasms; Neurotoxicity Syndromes | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): weekly chemotherapy
  Interventions: Drug: carboplatin; Drug: paclitaxel
- B (Active Comparator): every 3 weeks chemotherapy
  Interventions: Procedure: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Procedure: carboplatin — AUC 6 IV day 1 every 21 days
  Arms: B
Drug: paclitaxel — 175 mg/m2 IV day 1 every 21 days
  Arms: B
Drug: carboplatin — AUC 2 IV every week
  Arms: A
Drug: paclitaxel — 60mg/m2 IV every week
  Arms: A

SUMMARY:
The purpose of this study is to study efficacy and the effects on quality of life in women with ovarian cancer treated with a weekly schedule of chemotherapy with carboplatin and paclitaxel compared to those treated with standard every 3 weeks schedule of the same chemotherapy.

DETAILED DESCRIPTION:
The standard first-line treatment of ovarian cancer is combination chemotherapy with carboplatin and paclitaxel, given every 3 weeks. Researchers are looking at new ways of giving chemotherapy to make it more tolerable and more effective. One way is by giving the chemotherapy more often in smaller doses. This approach can be associated with fewer or less troubling side effects. Some chemotherapy drugs such as paclitaxel have been shown to also be more active when given once a week rather than once every 3 week schedule.

ELIGIBILITY:
Inclusion Criteria:

* Cytologic or histologic diagnosis of ovarian carcinoma of the ovary, fallopian tube or primary peritoneal carcinoma, stage IC-IV
* Indication for chemotherapy
* Age > 18 years
* Life expectancy of at least 3 months

Exclusion Criteria:

* Previous or concomitant malignant malignancy (excluding adequately treated baso-or squamocellular carcinoma of the skin and carcinoma in situ of the cervix, and synchronous endometrioid carcinoma Stage Ib or less for the uterus, with ovarian tumor Stage II or higher)
* Performance Status (ECOG) > or = 3.
* Previous chemotherapy
* Heart disease (congestive heart failure, myocardial infarction within 6 months from study entry, atrioventricular block of any grade, severe arrhythmias)
* Neutrophils < 2000 x mm3, platelets < 100000 x mm3
* Inadequate renal function (creatinine > or = 1.25 x normal values) or liver function (ALT or AST > or = 1.25 x normal values)
* Present or suspected hemorrhagic syndromes
* Inability to comply with protocol and follow-up
* Inability to access study site for clinical visits
* Refusal of informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2008-11 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
quality of life | weekly for the first 9 weeks of therapy, then every 3 weeks until the completion of therapy
progression free survival | every 6 months

SECONDARY OUTCOMES:
overall survival | 24 months
response rate | after 9 and 18 weeks of therapy
toxicity | weekly during therapy
describe the frequency and duration of symptoms in 12 months preceding ovarian cancer diagnosis | at study entry
describe time intervals of prediagnostic sentinel events (onset of persistent symptoms, first physician visit, diagnosis of ovarian cancer) | at study entry
describe patients' pathway to diagnosis of ovarian cancer according to modified Andersen's model of 'total patient delay' | at study entry

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Marilina Piccirillo, M.D.,, Principal Investigator — National Cancer Institute, Naples; Ciro Gallo, M.D., Ph.D., Principal Investigator — University of Campania Luigi Vanvitelli
Locations (28):
- Italy (28):
  - IRCCS Oncologico Bari, Oncologia Medica, Bari, BA
  - Ospedale Riuniti di Bergamo, U.O. di Ostetricia e Ginecologia, Bergamo, BG
  - Ospedale Fatebenefratelli, U.O. di Oncologia, Benevento, BN
  - Azienda Ospedaliera G. Rummo, Benevento, BN
  - Università Cattolica del Sacro Cuore, Dipartimento di Oncologia, Campobasso, CB
  - Azienda Ospedaliera C. Poma, Mantova, MN
  - Azienda Ospedaliera V. Cervello, Palermo, PA
  - Ospedale S. Massimo, Day Hospital Oncologico, Penne, PE
  - Centro di Riferimento Oncologico, Divisione di Oncolgia Medica C, Aviano, PN
  - Ospedale S. Chiara, Trento, TN
  - Ospedale S. Bortolo ULSS 6, U.O. di Oncologia Medica, Vicenza, VI
  - Ospedale Mazzoni, Ascoli Piceno
  - Policlinico Universitario, Bari
  - Universita di Bari Policinico I Clinical Ostetrica e Ginecologica, Bari
  - Ospedale Fatebenefratelli, Benevento
  - Ospedale Senatore Antonio Perrino, Brindisi
  - Universita Cattolica del Sacro Cuore, Campobasso
  - Ospedale A. Manzoni, Lecco
  - Istituto Nazionale Tumori, Milan
  - A.O. Univeristaria Policlinico, Modena
  - Azienda Ospedaliera D. Cotugno, Napoli
  - Istituto Nazionale dei Tumori , Oncologia Medica - Dipartimento Uro-Ginecologico, Napoli
  - Università Federico II, Cattedra di Oncologia Medica, Napoli
  - Ospedale Silvestrini, Perugia
  - Ospedale Civile S. Spirito, Pescara
  - A.O. S. Maria degli Angeli, Pordenone
  - Ospedale S. Giovanni Calibita Fatebenefratelli, UO di Oncologia, Roma
  - A.O. di Udine S. Maria della Misericordia, Udine

REFERENCES:
- [Result] Pignata S, Scambia G, Katsaros D, Gallo C, Pujade-Lauraine E, De Placido S, Bologna A, Weber B, Raspagliesi F, Panici PB, Cormio G, Sorio R, Cavazzini MG, Ferrandina G, Breda E, Murgia V, Sacco C, Cinieri S, Salutari V, Ricci C, Pisano C, Greggi S, Lauria R, Lorusso D, Marchetti C, Selvaggi L, Signoriello S, Piccirillo MC, Di Maio M, Perrone F; Multicentre Italian Trials in Ovarian cancer (MITO-7); Groupe d'Investigateurs Nationaux pour l'Etude des Cancers Ovariens et du sein (GINECO); Mario Negri Gynecologic Oncology (MaNGO); European Network of Gynaecological Oncological Trial Groups (ENGOT-OV-10); Gynecologic Cancer InterGroup (GCIG) Investigators. Carboplatin plus paclitaxel once a week versus every 3 weeks in patients with advanced ovarian cancer (MITO-7): a randomised, multicentre, open-label, phase 3 trial. Lancet Oncol. 2014 Apr;15(4):396-405. doi: 10.1016/S1470-2045(14)70049-X. Epub 2014 Feb 28. PMID 24582486